CLINICAL TRIAL: NCT01388049
Title: e- Ab Sensor - Based Real-time Diagnosis of Enterovirus Type 71
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: 201007053R
Record Dates: First submitted 2011-07-01; First posted 2011-07-06 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2011-11

CONDITIONS: EV71
Keywords: EV71

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- virus detection (Experimental)
  Interventions: Device: Electrosensing antibody probing system (e- Ab sensor)

INTERVENTIONS:
Device: Electrosensing antibody probing system (e- Ab sensor) — Electrosensing antibody probing system (e- Ab sensor), which was developed for the rapid and sensitive detection of hapten, proteins, or viral antigen in medical samples, will be used for analyzing the interaction kinetics between anti-EV71 antibody and its antigen (EV71) present in patients. The system incorporates the use of engineered semiconducive antibodies or virus in vertical and lateral chip (eAbchip) or lateral flow through (eAbsignal) formats. In electrosensing antibody probing, semiconductive antibodies are bound as a suitable electrosensing probe, which specifically and selectively binds targeted molecules (EV71) in the test specimens. From assessment of the electric signature of semiconductive anti-EV71 antibodies, the eABprobe could offer sensitive detection and precise quantification of EV71.

SUMMARY:
To develop a real-time diagnostic technique with e- Ab sensor for Entervirus 71 detection, the investigators conduct a prospective clinical study. In comparison with results from direct sequencing of Entervirus 71, the investigators evaluate the performance of e- Ab sensor, including reproducibility, sensitivity, specificity, and cross-reaction. The potential factors which may interfere with the results would be investigated. With such technique, the investigators hope to make early diagnosis and give EV71 patients early treatment to reduce the complications and case-fatality rate.

DETAILED DESCRIPTION:
Entervirus 71 is one of the most important infectious diseases in children and the important concern in public health. Since 1998, EV71 has become an endemic disease in Taiwan and caused hundreds of severe cases and dozens of fatal cases each year due to lack of EV71 vaccine. Family transmission study also showed that it is highly contagious among households as well as in daycares or kindergartens. Therefore, a rapid diagnosis is clinically necessary and can provide clinicians the rapid answers and make early treatment possible to reduce the complications and case-fatality rate. In addition, early diagnosis of the patients will alert parents and public health workers to prevent the contacts earlier and to limit the EV71 spread.

Electrosensing antibody probing system (e- Ab sensor), which was developed for the rapid and sensitive detection of hapten, proteins or viral antigen in medical samples, will be used for analyzing the interaction kinetics between Q.anti-EV71 and its antigen EV71 present in EV71 patients and normal sample. The system incorporates the use of engineered semiconductive antibodies or virus in vertical and lateral chip (eVchip) or lateral flow through (eVsignal) formats. In electrosensing virus probing, semiconductive antibodies are bound as a suitable electrosensing probe which specifically and selectively binds EV71 epitope target molecules in the test serum. In comparison with results from direct sequencing of EV71, the investigators evaluate the performance of e- Ab sensor, including reproducibility, sensitivity, specificity, and cross-reaction. The potential factors which may interfere with the results would be investigated. e- Ab sensor threshold decisions must maximize its sensitivity. Therefore, the threshold value in the test group is to find the decision could have 90% sensitivity and 90% specificity. With such technique, the investigators hope to make early diagnosis and give EV71 patients early treatment to reduce the complications and case-fatality rate.

ELIGIBILITY:
Inclusion Criteria:

* A: The patients with confirmed or suspected infection.
* B: The patients without disease.

Exclusion Criteria:

* Patients will be excluded if they couldn't sign the consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2010-07; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
The performance of e- Ab sensor | 1 Day
  In comparison with results from direct sequencing of EV71, we evaluate the performance of e- Ab sensor, including reproducibility, sensitivity, specificity, and cross-reaction.

CONTACTS AND LOCATIONS:
Overall Officials: Luan-Yin Chang, MD,PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan